CLINICAL TRIAL: NCT03911583
Title: Effectiveness of PUSH Notifications From a Mobile App for Improving the Body Composition of Overweight or Obese Women. Protocol of a Three-armed Clinical Assay
Brief Title: Effectiveness of PUSH Notifications From a Mobile App for Improving the Body Composition of Overweight or Obese Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidad de Córdoba (Other)
Responsible Party: Principal Investigator, Alberto Hernández de los Reyes, Principal Investigator, Universidad de Córdoba
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: V2-A284R4156
Record Dates: First submitted 2019-04-09; First posted 2019-04-11 (Actual); Last update posted 2019-04-11 (Actual); Status verified 2019-04

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — Control Groups

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (CG) (Active Comparator): Education, modifying diet and light physical activity (LPA)
  Interventions: Behavioral: Control Group (CG)
- Moderate physical activity group (MPA) (Active Comparator): Education, modifying diet and moderate physical activity (MPA)
  Interventions: Behavioral: Moderate physical activity group (MPA)
- Intense physical activity group (IPA) (Active Comparator): Education, modifying diet and intense physical activity (IPA)
  Interventions: Behavioral: Intense physical activity group (IPA)

INTERVENTIONS:
Behavioral: Control Group (CG) — The control group does not receive these notifications (PUSH)
  Arms: Control Group (CG)
Behavioral: Moderate physical activity group (MPA) — The women of the experimental group receive PUSH notifications remembering the objective set in consultation and encouraging them to achieve it.
  Arms: Moderate physical activity group (MPA)
Behavioral: Intense physical activity group (IPA) — The women of the experimental group receive PUSH notifications remembering the objective set in consultation and encouraging them to achieve it.
  Arms: Intense physical activity group (IPA)

SUMMARY:
A clinical three-armed assay has been established to permit an evaluation of the effectiveness of implementing PUSH notifications in the actions orientated towards improving body composition through the establishment of dietary patterns and an increase in physical activity.

DETAILED DESCRIPTION:
The use of mobile technology is already part of the investigator's daily life and its presence is increasing exponentially. The term mHealth (mobile health) was used and defined for the first time in 2000. This concept was subsequently employed in the 2010 mHealth Summit of the Foundation for National Institutes of Health (FNIH) to refer to "the provision of medical attention services through mobile communication devices". Around 40% of the over 300,000 applications available in the different apps stores are related to health themes, with those focused on the monitoring and management of diseases standing out. One of the characteristics of mobile applications is the sending and receiving of messages through a system of notifications known as "PUSH", that consists of requests appearing on the display of the Smartphone at a scheduled time, permitting them to be customizable both in their contents and at the time of sending them

PUSH notifications are pro-active as they offer visual and/or aural alerts to inform the recipient of a message or event received and invite them to act on them, even without the App being in use. On receiving the notification, the user can interact in different degrees, from simply reading it to answering it, thus permitting feedback. Also, there is evidence of the PUSH notifications being effective in communications between professionals.

The objective of this study is to compare the effect of the implementation of a monitoring system, goal to achieve, on physical activity in overweight and obese adults. A clinical three-armed assay has been established to permit an evaluation of the effectiveness of implementing PUSH notifications in the actions orientated towards improving body composition through the establishment of dietary patterns and an increase in physical activity.

Participants (n=90) will be recruited through outpatient from private clinics in Cádiz, Andalucía, Spain, as well as through community presentations. Overweight or obese and sedentary adult will be randomly assigned into three groups.

For 6 months, all of the adults shall follow the same diet with an identical distribution of macronutrients. There will be a weekly check up of weight, fat, body water and muscle mass for all of them. The status of the number of steps in Accupedo is also checked every week.

ELIGIBILITY:
Inclusion Criteria:

* Having a IMC >25,
* Being sedentary and
* Have not been submitted to a restrictive diet in the 6 months preceding this study.
* Having a body fat percentage of ≥ 30%

Exclusion Criteria:

* Suffered from type 2 diabetes or renal conditions
* Being pregnancy or attempt at pregnancy,
* Being in a maternal lactation period,
* Not possessing a Smartphone with an operating system (Android or iOS) and available data connection did not participate in the study.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 90 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-12-15 (Actual); Study Completion 2019-06-01 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline BMI | At baseline (0 years) and followed for 2 years
  Baseline mean BMI values will be measured and compared at 3, 6, 12 and 24 months. BMI will be assessed on a monthly basis during nutritional consultation through a Bioelectrical Impedance Analysis method using a Tanita BC-418 Segmental Body Composition Analyser/Scale
Changes from baseline Fatty mass | At baseline (0 years) and followed for 2 years
  Baseline mean Fatty mass values will be measured and compared at 3, 6, 12 and 24 months. Fatty mass will be assessed on a monthly basis during nutritional consultation through a Bioelectrical Impedance Analysis method using a Tanita BC-418 Segmental Body Composition Analyser/Scale. Fatty mass is measured as a percentage.
Changes from baseline Free-fatty mass | At baseline (0 years) and followed for 2 years
  Baseline mean Free-fatty mass values will be measured and compared at 3, 6, 12 and 24 months. Free-fatty mass will be assessed on a monthly basis during nutritional consultation through a Bioelectrical Impedance Analysis method using a Tanita BC-418 Segmental Body Composition Analyser/Scale. Fatty mass is measured as a percentage.
Changes from baseline Muscular Mass | At baseline (0 years) and followed for 2 years
  Baseline mean Muscular Mass values will be measured and compared at 3, 6, 12 and 24 months. Muscular Mass will be assessed on a monthly basis during nutritional consultation through a Bioelectrical Impedance Analysis method using a Tanita BC-418 Segmental Body Composition Analyser/Scale. Fatty mass is measured as a Kg.
Changes from baseline Corporal Water | At baseline (0 years) and followed for 2 years
  Baseline mean Corporal Water values will be measured and compared at 3, 6, 12 and 24 months. Corporal Water will be assessed on a monthly basis during nutritional consultation through a Bioelectrical Impedance Analysis method using a Tanita BC-418 Segmental Body Composition Analyser/Scale. Fatty mass is measured as a Kg.
Adherence to dietary pattern will be also measured through personal interview | At baseline (0 years) and followed for 2 years
  Participants will be subjected for an intervention based on nutritional (control group) and physical education (two intervention arms) during 24 months. Partial measures will be also taken every week. In the end of the trial, changes in dietary patterns will be measured comparing means differences between baselines, 3, 6, 12 and 24 months.
Adherence to physical activity patterns will be also measured through IPAQ (International Physical Activity Questionnaire) | At baseline (0 years) and followed for 2 years
  Participants will be subjected for an intervention based on nutritional (control group) and physical education (two intervention arms) during 24 months. Partial measures will be also taken every week. In the end of the trial, changes in physical activity will be measured comparing means differences between baselines, 3, 6, 12 and 24 months.

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Hernández-Reyes, M.Sc., Principal Investigator — Universidad de Córdoba

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hernandez-Reyes A, Molina-Recio G, Molina-Luque R, Romero-Saldana M, Camara-Martos F, Moreno-Rojas R. Effectiveness of PUSH notifications from a mobile app for improving the body composition of overweight or obese women: a protocol of a three-armed randomized controlled trial. BMC Med Inform Decis Mak. 2020 Feb 24;20(1):40. doi: 10.1186/s12911-020-1058-7. PMID 32093701
- [Derived] Hernandez-Reyes A, Camara-Martos F, Molina Recio G, Molina-Luque R, Romero-Saldana M, Moreno Rojas R. Push Notifications From a Mobile App to Improve the Body Composition of Overweight or Obese Women: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2020 Feb 12;8(2):e13747. doi: 10.2196/13747. PMID 32049065